CLINICAL TRIAL: NCT00351507
Title: A Double-blind, Crossover, Placebo-Controlled, Multiple-dose Study to Evaluate the Effects of Vildagliptin on Gastric Emptying, Gastric Volume and Satiety in Patients With Type 2 Diabetes
Brief Title: A Study to Assess the Effects of Vildagliptin on Gastric Emptying in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2343
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Vildagliptin; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin

SUMMARY:
This study was designed to directly assess the effects of vildagliptin on gastric emptying in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for at least 6 months
* Blood glucose criteria must be met
* BMI in the range 22-40

Exclusion Criteria:

* History of type 1 diabetes, diabetes resulting from pancreatic injury, or secondary forms of diabetes
* Use of thiazolidinediones or need for insulin within 3 months prior to screening
* Significant concomitant diseases or complications of diabetes
* High fasting triglycerides as defined by the protocol

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-05; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Effect on gastric emptying

SECONDARY OUTCOMES:
Effect on gastric volume
Effect on satiety
Effect on endogenous glucose appearance, glucose appearance and glucose disposal

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic & Foundation
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Dalla Man C, Bock G, Giesler PD, Serra DB, Ligueros Saylan M, Foley JE, Camilleri M, Toffolo G, Cobelli C, Rizza RA, Vella A. Dipeptidyl peptidase-4 inhibition by vildagliptin and the effect on insulin secretion and action in response to meal ingestion in type 2 diabetes. Diabetes Care. 2009 Jan;32(1):14-8. doi: 10.2337/dc08-1512. Epub 2008 Oct 17. PMID 18931099